CLINICAL TRIAL: NCT02474147
Title: Effects of Processed Meat on Brain Regions Related to Reward and Craving in Patients With Type 2 Diabetes, Obese Subjects and Healthy Controls
Brief Title: Processed Meat and Brain Regions Related to Reward and Addiction
Acronym: RewCrav
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Hana Kahleova, MD, PhD, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: G251
Record Dates: First submitted 2015-06-02; First posted 2015-06-17 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Type 2 diabetics (Experimental): Patients with type 2 diabetes Interventions: processed meat hamburger and vegan sandwich
  Interventions: Other: Processed meat hamburger; Other: Vegan sandwich
- Obese subjects (Active Comparator): Obese subjects without diabetes Interventions: processed meat hamburger and vegan sandwich
  Interventions: Other: Processed meat hamburger; Other: Vegan sandwich
- Healthy lean controls (Active Comparator): Healthy lean controls Interventions: processed meat hamburger and vegan sandwich
  Interventions: Other: Processed meat hamburger; Other: Vegan sandwich

INTERVENTIONS:
Other: Processed meat hamburger — MacMuffin Fresh 300 ml Cafe Latte + 21 g sugar Energy: 513.6 kcal Carbohydrates 55g (44.8%) Proteins 20.5g (16.7%) Lipids 22 g (38.6%)
Other: Vegan sandwich — Burger with tofu + 300 ml green tea Energy 514.9 kcal Carbohydrates 54.2 g (44%) Proteins 19.9 g (16.2%) Lipids 22.8 g (39.8%)

SUMMARY:
The purpose of this study is to

1. Compare effects of two isocaloric meals (processed meat hamburger vs. vegetarian sandwich) in response to the postprandial period by using functional brain imaging of reward circuitry implicated in food motivation and energy balance in patients with type 2 diabetes (T2D), obese subjects and healthy controls.
2. Characterize some of the pathophysiological mechanisms of action of different meals in obese and T2D subjects vs. in healthy controls (serum concentrations of glucose, FFA, IRI, C-peptide, gastrointestinal hormones, oxidative stress markers)

DETAILED DESCRIPTION:
The mesolimbic dopaminergic system of the brain, which converges on the nucleus accumbens (part of the striatum), plays a central role in reward and craving, and this system appears to mediate hedonic food responses. In rodent studies, extracellular concentrations of dopamine and its metabolites in the nucleus accumbens increased more after the consumption of highly palatable food than standard rodent feed pellets. Furthermore, microinjections of opiate into the nucleus accumbens increased food intake and the reward value of food. Clinical studies that used functional brain imaging have reported greater activation in the nucleus accumbens or other regions of the striatum in obese than lean individuals after they viewed or consumed palatable, high-calorie food. Of particular interest, striatal dopamine D2 receptor availability was significantly lower in obese individuals than in nonobese matched controls, which raised the possibility that overeating may compensate for low dopaminergic activity. The recurrent activation of the striatum may down-regulate dopamine availability and further heighten the drive to overeat. However, the information on the exact effect of different foods and nutrients on the mesolimbic dopaminergic system is missing.

Preliminary findings that lead to the project

A positive association between high consumption of total and red meat, especially processed meat, and incidence of T2D has been demonstrated. Previous studies support the concept that increased oxidative stress may play an important role in T2D manifestation. Dietary fat quality has been proposed to be a critical factor. Several studies have suggested that a high intake of saturated fatty acids naturally present in meat contributes to the risk of glucose intolerance. In an intervention study, humans suffering from metabolic syndrome who were consuming a diet rich in saturated fats displayed higher oxidative stress markers postprandially. It is not clear if saturated fatty acids per se or via increased oxidative stress markers may activate the mesolimbic dopaminergic system.

In contrast, some intervention trials (including ours) demonstrated a greater improvement in insulin sensitivity, glycemic control and a reduction in oxidative stress markers in T2D patients consuming a vegetarian diet compared to a conventional diabetic diet. The effect of a vegetarian diet on the mesolimbic dopaminergic system has not been studied yet.

Aims and priorities of the project

The purpose of this study is to

1. Compare effects of two isocaloric meals (processed meat hamburger vs. vegetarian sandwich) in response to the postprandial period by using functional brain imaging of reward circuitry implicated in food motivation and energy balance in patients with type 2 diabetes (T2D), obese subjects and healthy controls.
2. Characterize some of the pathophysiological mechanisms of action of different meals in obese and T2D subjects vs. in healthy controls (serum concentrations of glucose, FFA, IRI, C-peptide, gastrointestinal hormones, oxidative stress markers)

Hypothesis

1. Obese and T2D subjects relative to lean healthy controls will show greater activation in the gustatory cortex and in somatosensory regions in response to the intake of processed meat hamburger (vs. a vegetarian sandwich). However, they will also show decreased activation in the caudate nucleus in response to consumption of processed meat hamburger (vs. a vegetarian sandwich).
2. Changes in serum concentrations of glucose, FFA, IRI, C-peptide, gastrointestinal hormones and oxidative stress markers will be involved in gut-brain axis signaling. The investigators hypothesise to find an association between postprandial changes in serum concentrations of FFA and postprandial changes in activation in the gustatory cortex and in somatosensory regions of the brain.

The actual need for this study The pandemic of obesity and diabetes especially in western countries calls for high-quality research and relevant action. A better understanding of the pathophysiological mechanisms of the stimulation of brain regions involved in reward and craving in response to processed meat, one of the most significant present risk factors for obesity and type 2 diabetes, is needed in order to develop more effective preventive and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for T2D:

1. Type 2 diabetes mellitus for at least one year
2. Treatment of T2D: diet or oral antidiabetic agents (stable drug therapy at least 3 month before the trial
3. The presence of metabolic syndrome - any three of the following symptoms:

   * Abdominal obesity - waist circumf. in men> 102 cm, in women > 88 cm
   * Diagnosis and treatment of type 2 diabetes or raised fasting plasma glucose level (FPG>5,6 mmol/l)
   * Raised blood pressure (BP): systolic BP > 130 mm Hg or diastolic BP >85 mm Hg, or treatment of previously diagnosed hypertension
   * Reduced HDL cholesterol in men < 1 mmol/l, in women < 1,3 mmol/l (or treatment)
   * Raised triglycerides > 1,7 mmol/l (or treatment)
4. HbA1c (according to IFCC) ≥4.2 a ≤10.5%
5. Men and women aged 30-70 years
6. Body Mass Index (kg/m2) in the range of 25- 45
7. The signed informed consent

Exclusion Criteria:

Exclusion criteria for T2D:

1. Type 1 diabetes mellitus
2. Unstable drug therapy at least 3 month before the trial
3. Treatment with Byetta or Victosa
4. Pregnancy (positive β-HCG test), breast feeding or trying to become pregnant
5. Presence of pacemaker or other metal implant in the body (MR)
6. Alcoholism or drug use
7. Significant weight loss (more than 5% of body weight) in previous 3 months before the screening
8. Presence of other medical condition, which occurs during physical examination, laboratory tests, ECG, including pulmonary, neurological or inflammatory disease, which would be considered by the examiner to distort the consistency of data
9. Metal in the body (fMRI)

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Functional brain imaging of reward circuitry | 24 months
  fMRI (functional magnetic resonance imaging) of the brain pre- and postprandially simultaneously with both meal tests with the use of the modern method of arterial spin labeling (ASL) which allows quantification of the blood perfusion of the brain regions involved in craving and reward.

SECONDARY OUTCOMES:
Serum concentrations of gastrointestinal hormones | 24 months
  Plasma concentrations of selected gut hormones will be measured enzymatically using standard kits
Serum concentrations of oxidative stress markers | 24 months
  Plasma concentrations of selected oxidative stress markers will be measured enzymatically using standard kits

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Koveslygetyova, Bc, Study Chair — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czech Republic, Czechia

REFERENCES:
- [Derived] Malinska H, Klementova M, Kudlackova M, Veleba J, Hoskova E, Oliyarnyk O, Markova I, Thieme L, Hill M, Pelikanova T, Kahleova H. A plant-based meal reduces postprandial oxidative and dicarbonyl stress in men with diabetes or obesity compared with an energy- and macronutrient-matched conventional meal in a randomized crossover study. Nutr Metab (Lond). 2021 Sep 10;18(1):84. doi: 10.1186/s12986-021-00609-5. PMID 34507586
- [Derived] Kahleova H, Tintera J, Thieme L, Veleba J, Klementova M, Kudlackova M, Malinska H, Oliyarnyk O, Markova I, Haluzik M, Pavlovicova R, Hill M, Tura A, Pelikanova T. A plant-based meal affects thalamus perfusion differently than an energy- and macronutrient-matched conventional meal in men with type 2 diabetes, overweight/obese, and healthy men: A three-group randomized crossover study. Clin Nutr. 2021 Apr;40(4):1822-1833. doi: 10.1016/j.clnu.2020.10.005. Epub 2020 Oct 9. PMID 33081982